CLINICAL TRIAL: NCT00868010
Title: Donepezil to Promote Functional Recovery Post-stroke
Brief Title: Enhancing Rehabilitation After Stroke
Acronym: Enhance
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Ellen Whyte, Principal Investigator, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R01HD055525 (NIH); NIH grant: 1 R01 HD055525-01A2
Record Dates: First submitted 2009-03-22; First posted 2009-03-24 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Ischemic Stroke
Keywords: stroke; donepezil; recovery
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1: donepezil (Experimental): Participants will receive treatment for 12 weeks on donepezil 10 mg (or 5 mg if unable to tolerate 10 mg). Treatment will be then be terminated and participants followed for another 12 weeks naturalistically.
  Interventions: Drug: donepezil
- 2. placebo (Placebo Comparator): Participants will receive treatment for 12 weeks with placebo pill. Treatment will be then be terminated and participants followed for another 12 weeks naturalistically.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: donepezil — 5 mg or 10 mg, titrated per drug insert. Participants may remain in the study at 5 mg if unable to tolerate 10 mg.
  Other Names: Aricept
  Arms: 1: donepezil
Drug: placebo — Participants will receive a placebo pill for 12 weeks if randomized to this treatment.
  Arms: 2. placebo

SUMMARY:
This is a 12-week, randomized, placebo controlled study to determine if donepezil (Aricept) treatment during rehabilitation after stroke improves functional recovery.

DETAILED DESCRIPTION:
Stroke is a leading cause of disability in the US (Thom 2006). The total number of stroke survivors (currently estimated as 5.5 million Americans) will continue to increase as the population ages and as the medical management of acute stroke continues to improve. Given stroke's devastating impact on activities of daily living and the large numbers of Americans afflicted, improving acute medical rehabilitation outcomes after stroke is of great public health importance.

Predictors of poor functional recovery post-stroke include impairments in cognition and motivation. Recent evidence indicates that acetylcholinesterase inhibitors may improve cognition and motivation; hence, their use post-stroke may lead to improved rehabilitation outcomes. Our group has demonstrated that use of the acetylcholinesterase inhibitor donepezil is associated with improved functional recovery in a pilot sample (n = 40) of elderly, cognitively impaired stroke survivors undergoing inpatient rehabilitation. Specifically, in this 12 week open-label study, those subjects receiving donepezil experienced a clinically meaningful 14 point greater improvement on the Functional Independence Measure (FIM) than an archival comparator group.

Based on these promising pilot study results, we propose a 12-week randomized, double-blind, placebo-controlled trial (followed by a 12 week off-drug observation period) in order to test the efficacy of donepezil to promote post-stroke functional recovery in older, cognitively impaired stroke survivors undergoing inpatient rehabilitation. We will also use this randomized controlled trial to examine the drug's effect on cognition post-stroke; specifically, the drug's effect on those cognitive domains (attention/working memory, information psychomotor speed, and episodic memory) that are relevant to functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. male or female;
2. aged 18 or older;
3. new ischemic stroke within the preceding 30 days; and
4. admitted to the an inpatient facility of the UPMC Institute for Rehabilitation and Research for post-stroke rehabilitation.

Exclusion Criteria:

1. primary hemorrhagic stroke;
2. current use of a cholinomimetic drug including tacrine, donepezil, galantamine, and rivastigmine;
3. contraindication to AchEi therapy including bradycardia (< 50 bpm), severe asthma or COPD requiring nebulized medication, and active upper GI bleed or untreated gastric ulcer;
4. myocardial infarction, poorly controlled congestive heart failure, or coronary bypass surgery within the last 3 months;
5. current required use of an anticholinergic medication (e.g., for bladder spasm);
6. current aphasia severe enough to prevent valid neuropsychiatric assessment (e.g., a score < 9 on the Token Test, part I and a score of < 14 (or <80% accuracy) on the repetition task of the Boston Diagnostic Aphasia Examination);
7. current Major Depressive Episode AND HRSD > 20;
8. current active suicidal ideation, plan, or intent;
9. current mania or hypomania;
10. current psychosis;
11. meeting DMS-IV TR alcohol or substance abuse or dependence criteria within the preceding 3 months;
12. subject and/or family informant do not speak English;
13. history of a progressive or unstable CNS disease (e.g., multiple sclerosis, Parkinson's disease, HIV with CNS involvement);
14. medically unstable (determined by review of the subject's medical status with the treating (clinical) physician and by review of standard blood tests); and
15. history of sensitivity to donepezil;
16. for potential subjects without a pacemaker or implantable defibrillator, exclusion criteria will include (a) ECG evidence of second or third degree heart block ( b ) ECG evidence of a tri-fascicular block (LBBB and 1st degree AV Block; RBBB, left anterior or left posterior hemiblock, and 1st degree AV block) or ( c ) history of syncope within 1 year with a RBBB or a LBBB.
17. For females of child-bearing age, current pregnancy, plan to become pregnant while on study drug, or refusal to avoid pregnancy while on study drug.
18. For females of child-bearing age, current breast feeding.
19. suicidal attempt in the past one year,
20. an inpatient admission for depression in the past one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-03; Primary Completion 2013-08 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Functional Independence Measure (FIM) | Weekly/12 weeks

SECONDARY OUTCOMES:
Cognitive Function (ImPACT battery used to assess attention - working memory continuum, information processing speed, and verbal and visual episodic memory.) | Multiple time points over 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ellen M Whyte, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Hillside Rehabilitation Hospital, Warren, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Thom T, Haase N, Rosamond W, Howard VJ, Rumsfeld J, Manolio T, Zheng ZJ, Flegal K, O'Donnell C, Kittner S, Lloyd-Jones D, Goff DC Jr, Hong Y, Adams R, Friday G, Furie K, Gorelick P, Kissela B, Marler J, Meigs J, Roger V, Sidney S, Sorlie P, Steinberger J, Wasserthiel-Smoller S, Wilson M, Wolf P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2006 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2006 Feb 14;113(6):e85-151. doi: 10.1161/CIRCULATIONAHA.105.171600. Epub 2006 Jan 11. No abstract available. PMID 16407573
- [Background] Whyte EM, Lenze EJ, Butters M, Skidmore E, Koenig K, Dew MA, Penrod L, Mulsant BH, Pollock BG, Cabacungan L, Reynolds CF 3rd, Munin MC. An open-label pilot study of acetylcholinesterase inhibitors to promote functional recovery in elderly cognitively impaired stroke patients. Cerebrovasc Dis. 2008;26(3):317-21. doi: 10.1159/000149580. Epub 2008 Jul 31. PMID 18667813
- See also: American Stroke Association website provides general information regarding stroke and stroke prevention. — http://www.strokeassociation.org